CLINICAL TRIAL: NCT00391391
Title: Immunogenicity and Safety of a Split, Inactivated, Trivalent Influenza Vaccine Administered by Intradermal Route in Comparison With Intramuscular Vaccination With Standard Fluzone® in Healthy Infants and Young Children.
Brief Title: Study of Inactivated, Split-Virion Influenza Vaccine Compared With Standard Fluzone Vaccine in Infants and Children
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: FID07
Record Dates: First submitted 2006-10-23; First posted 2006-10-24 (Estimated); Results first posted 2011-11-22 (Estimated); Last update posted 2011-12-01 (Estimated); Status verified 2011-11

CONDITIONS: Orthomyxoviridae Infection; Influenza; Myxovirus Infection
Keywords: Influenza; Orthomyxoviruses; Inactivated Split-virion influenza vaccine; Infants; children.
MeSH Terms: conditions — Orthomyxoviridae Infections; Influenza, Human | interventions — Influenza Vaccines

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- 1 (Experimental): Split, Inactivated, Trivalent Influenza Vaccine
  Interventions: Biological: Split, Inactivated, Trivalent Influenza Vaccine
- 2 (Experimental): Split, Inactivated, Trivalent Influenza Vaccine
  Interventions: Biological: Split, Inactivated, Trivalent Influenza Vaccine
- 3 (Active Comparator): Split, Inactivated, Trivalent Influenza Vaccine
  Interventions: Biological: Split, Inactivated, Trivalent Influenza Vaccine ( Fluzone® 2006/2007 Formulation)
- 4 (Active Comparator): Split, Inactivated, Trivalent Influenza Vaccine
  Interventions: Biological: Split, Inactivated, Trivalent Influenza Vaccine ( Fluzone® 2006/2007 Formulation)

INTERVENTIONS:
Biological: Split, Inactivated, Trivalent Influenza Vaccine — Vaccine (infant dose)
  Arms: 1
Biological: Split, Inactivated, Trivalent Influenza Vaccine — Vaccine (children dose)
  Arms: 2
Biological: Split, Inactivated, Trivalent Influenza Vaccine ( Fluzone® 2006/2007 Formulation) — Vaccine (infant dose)
  Other Names: Fluzone® 2006/2007 Formulation.
  Arms: 3
Biological: Split, Inactivated, Trivalent Influenza Vaccine ( Fluzone® 2006/2007 Formulation) — Vaccine (children dose)
  Other Names: Fluzone® 2006/2007 Formulation.
  Arms: 4

SUMMARY:
Primary Objective:

To evaluate for each influenza strain the non-inferiority of Investigational Fluzone vaccine to the standard Fluzone® vaccine in healthy subjects aged 6 to 35 months or 3 to 8 years.

Secondary Objectives:

* To describe the immunogenicity of of Investigational Fluzone vaccine to the standard Fluzone® vaccine in healthy subjects aged 6 to 35 months or 3 to 8 years.
* To describe the safety of of Investigational Fluzone vaccine to the standard Fluzone® vaccine in healthy subjects aged 6 to 35 months or 3 to 8 years.

ELIGIBILITY:
Inclusion Criteria :

* Aged 6 months to 8 years but not yet 9 years on the day of inclusion.
* Subject is healthy, as determined by medical history.
* Institution Review Board (IRB)-approved informed assent form signed by eligible subject (if required by local regulations) and/or an IRB-approved informed consent form signed by the subject's parent(s) or legal representative (and by an independent witness if required by local regulations).
* Parent or legal guardian willing and able to attend (bring subject) to all scheduled visits and comply with all trial procedures.

Exclusion Criteria :

* Participation in another clinical trial in the 4 weeks preceding the trial vaccination.
* Planned participation in another clinical trial during the present trial period.
* Personal or family history of Guillain-Barré Syndrome.
* Congenital or acquired immunodeficiency, immunosuppressive therapy such as anti-cancer chemotherapy or radiation therapy within the preceding 6 months, or long-term systemic corticosteroid therapy injected or oral corticosteroids or other immunomodulator therapy within six weeks of the study vaccine. Individuals on a tapering dose schedule of oral steroids lasting < 7 days may be included in the trial as long as they have not received more than one course within the last two weeks prior to enrollment.
* Systemic hypersensitivity to eggs, chicken proteins, or any of the vaccine components, or a vaccine containing the same substances.
* Chronic illness at a stage that could interfere with trial conduct or completion
* Received blood or blood-derived products in the previous 3 months.
* Any vaccination in the 4 weeks preceding or following the trial vaccinations (Subjects can take standard childhood vaccination(s) following Visit 3 blood draw).
* Known current human immunodeficiency virus (HIV), hepatitis B (HBsAg) or hepatitis C infection or seropositivity.
* Known thrombocytopenia or bleeding disorder contraindicating IM vaccination.
* Acute medical illness, with or without fever, within the last 72 hours or an oral temperature ≥ 37.5 °C (99.5 °F) or rectal temperature of ≥ 38°C (100.4 °F) at the time of enrollment.
* History of seizures.
* Received antibiotics therapy within 72 hours preceding the trial vaccination.
* Received any allergy shots in the 7-day period preceding trial vaccination and/or scheduled to receive any allergy shots in the 7-day period after trial vaccination.
* Any condition, which in the opinion of the investigator would pose a health risk to the participant.

Ages: 6 Months to 8 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 520 (Actual)
Dates: Start 2006-10; Primary Completion 2007-03 (Actual); Study Completion 2007-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Sanofi Pasteur Inc.
Locations (18):
- United States (18):
  - Harrisburg, Arkansas
  - Little Rock, Arkansas
  - Trumann, Arkansas
  - Bellflower, California
  - Downey, California
  - Fountain Valley, California
  - Paramount, California
  - Owensboro, Kentucky
  - Bossier City, Louisiana
  - Shreveport, Louisiana
  - Brainerd, Minnesota
  - Cleveland, Ohio
  - Erie, Pennsylvania
  - Pittsburgh, Pennsylvania
  - Uniontown, Pennsylvania
  - Wexford, Pennsylvania
  - Fort Worth, Texas
  - Salt Lake City, Utah

REFERENCES:
- See also: Related Info — http://www.sanofipasteur.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study participants ere enrolled from 19 October to 12 December 2006 in 20 clinical centers in the US.
Pre-assignment Details: A total of 517 of the 520 participants who met the inclusion and exclusion criteria were enrolled and vaccinated.
Groups:
- Group 1: Fluzone ID at Age 6 to 35 Months: Participants at 6 to 35 Months of age on enrollment that received Fluzone ID vaccine
- Group 2: Fluzone IM 6 to 35 Months Age Group: Participants at 6 to 35 Months Age on enrollment that received Fluzone IM vaccine
- Group 3: Fluzone ID at 3 to 8 Years Age: Participants at Age 3 to 8 Years on enrollment that received Fluzone ID vaccine
- Group 4: Fluzone IM 3 to 8 Years Age: Participants at age 3 to 8 years on enrollment that received Fluzone IM vaccine
Period: Overall Study
Arm/Group | Group 1: Fluzone ID at Age 6 to 35 Months | Group 2: Fluzone IM 6 to 35 Months Age Group | Group 3: Fluzone ID at 3 to 8 Years Age | Group 4: Fluzone IM 3 to 8 Years Age
Started | 98 (1 participant was not vaccinated.) | 97 | 161 (1 participant was not vaccinated.) | 164 (1 participant was not vaccinated.)
Completed | 89 | 87 | 138 | 145
Not Completed | 9 | 10 | 23 | 19
Not completed — Adverse Event | 0 | 0 | 0 | 1
Not completed — Lost to Follow-up | 1 | 3 | 7 | 4
Not completed — Protocol Violation | 2 | 3 | 6 | 7
Not completed — Withdrawal by Subject | 6 | 4 | 10 | 7

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Group 1: Fluzone ID at Age 6 to 35 Months | Group 2: Fluzone IM 6 to 35 Months Age Group | Group 3: Fluzone ID at 3 to 8 Years Age | Group 4: Fluzone IM 3 to 8 Years Age | Total
Number analyzed (Participants) | 97 | 97 | 160 | 163 | 517
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 97 | 97 | 160 | 163 | 517
  Between 18 and 65 years | 0 | 0 | 0 | 0 | 0
  >=65 years | 0 | 0 | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: Months] | 22.6 (7.51) | 21.8 (8.03) | 69.6 (22.2) | 70.8 (21.6) | 46.5 (14.835)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 45 | 43 | 70 | 84 | 242
  Male | 52 | 54 | 90 | 79 | 275
Region of Enrollment [Number; unit: Participants]
  United States | 97 | 97 | 160 | 163 | 517

OUTCOME MEASURES:

1. Primary Outcome: Geometric Mean Titers (GMTs) Before and Post Vaccination With Either a Fluzone Intradermal or a Fluzone Intramuscular Vaccine
Description: Antibody titers against each strain of influenza hemagglutinin were measured in the sera using the hemagglutination inhibition (HI) technique.
Time Frame: Day 0 and Day 28 post-vaccination
Population: Geometric Mean Titers were determined in the per-protocol population.
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | Group 1: Fluzone ID at Age 6 to 35 Months | Group 2: Fluzone IM 6 to 35 Months Age Group | Group 3: Fluzone ID at 3 to 8 Years Age | Group 4: Fluzone IM 3 to 8 Years Age
Number analyzed (Participants) | 69 | 68 | 115 | 120
Titers
  Serogroup A/H1N1 Pre-vaccination | 8.9 [7.1 to 11.2] | 9.6 [7.5 to 12.3] | 20.5 [15.6 to 26.9] | 26.9 [19.6 to 37.1]
  Serogroup A/H1N1 Post-vaccination 1 | 58.5 [28.6 to 119.4] | 113.1 [59.9 to 213.7] | 100.1 [55.0 to 182.1] | 264.2 [162.8 to 428.9]
  Serogroup A/H1N1 Post-vaccination 2 | 138.3 [105.2 to 181.8] | 160.0 [123.7 to 206.9] | 162.9 [128.7 to 206.3] | 390.6 [308.2 to 495.0]
  Serogroup A/H3N2 Pre-vaccination | 22.4 [14.0 to 35.9] | 20.9 [13.7 to 31.9] | 222.2 [165.4 to 298.5] | 171.0 [121.5 to 240.7]
  Serogroup A/H3N2 Post-vaccination 1 | 341.8 [142.9 to 817.7] | 566.9 [304.6 to 1054.9] | 1012.5 [666.9 to 1537.2] | 1256.9 [898.2 to 1758.8]
  Serogroup A/H3N2 Post-vaccination 2 | 614.8 [471.3 to 802.0] | 471.4 [368.0 to 603.7] | 1111.0 [944.0 to 1307.5] | 1344.4 [1146.1 to 1577.1]
  Serogroup B Pre-vaccination | 5.3 [4.9 to 5.8] | 5.4 [5.0 to 5.9] | 8.3 [7.1 to 9.7] | 6.8 [6.0 to 7.7]
  Serogroup B Post-vaccination 1 | 7.4 [4.4 to 12.5] | 9.7 [4.2 to 22.1] | 46.6 [23.3 to 93.3] | 28.8 [16.0 to 52.0]
  Serogroup B Post-vaccination 2 | 31.1 [23.7 to 40.8] | 18.2 [13.9 to 24.0] | 56.4 [43.8 to 72.7] | 51.6 [40.8 to 65.2]

2. Secondary Outcome: Percentage of Participants That Achieved A 4-Fold Rise in Serum HAI Antibody Titer Post-vaccination With Either a Fluzone Intradermal or a Fluzone Intramuscular Vaccine
Description: as for outcome 1
Time Frame: Day 28 post-vaccination
Population: 4-Fold Rise in Serum HAI Antibody Titers were determined in the per-protocol population
Measure: Number; unit: Percentage of Participants
Arm/Group | Group 1: Fluzone ID at Age 6 to 35 Months | Group 2: Fluzone IM 6 to 35 Months Age Group | Group 3: Fluzone ID at 3 to 8 Years Age | Group 4: Fluzone IM 3 to 8 Years Age
Number analyzed (Participants) | 69 | 68 | 115 | 120
Percentage of Participants
  Serogroup A/H1N1 Post-vaccination 1 | 52 | 75 [0 to 0] | 65 [0 to 0] | 74 [0 to 0]
  Serogroup A/H1N1 Post-vaccination 2 | 91 | 88 [0 to 0] | 70 [0 to 0] | 78 [0 to 0]
  Serogroup A/H3N2 Post-vaccination 1 | 81 | 80 [0 to 0] | 44 [0 to 0] | 63 [0 to 0]
  Serogroup A/H3N2 Post-vaccination 2 | 88 | 91 [0 to 0] | 50 [0 to 0] | 62 [0 to 0]
  Serogroup B Post-vaccination 1 | 5 | 10 [0 to 0] | 44 [0 to 0] | 40 [0 to 0]
  Serogroup B Post-vaccination 2 | 44 | 21 [0 to 0] | 55 [0 to 0] | 53 [0 to 0]

3. Secondary Outcome: Percentage of Participants That Achieved Seroprotection Before and Post-vaccination With Either a Fluzone Intradermal or a Fluzone Intramuscular Vaccine
Description: Seroprotection was defined as participants achieving a post-dose antibody titers ≥40.
  Antibody titers against each strain of influenza hemagglutinin were measured in the sera using the hemagglutination inhibition (HI) technique.
Time Frame: Day 28 post-vaccination
Population: Seroprotection to vaccine antigens were determined in the per-protocol population
Measure: Number; unit: Percentage of Participants
Arm/Group | Group 1: Fluzone ID at Age 6 to 35 Months | Group 2: Fluzone IM 6 to 35 Months Age Group | Group 3: Fluzone ID at 3 to 8 Years Age | Group 4: Fluzone IM 3 to 8 Years Age
Number analyzed (Participants) | 69 | 68 | 115 | 120
Percentage of Participants
  Serogroup A/H1N1 Pre-vaccination | 9 | 12 [0 to 0] | 33 [0 to 0] | 40 [0 to 0]
  Serogroup A/H1N1 Post-vaccination 1 | 52 | 75 [0 to 0] | 79 [0 to 0] | 95 [0 to 0]
  Serogroup A/H1N1 Post-vaccination 2 | 91 | 93 [0 to 0] | 92 [0 to 0] | 99 [0 to 0]
  Serogroup A/H3N2 Pre-vaccination | 32 | 29 [0 to 0] | 86 [0 to 0] | 80 [0 to 0]
  Serogroup A/H3N2 Post-vaccination 1 | 85 | 95 [0 to 0] | 97 [0 to 0] | 100 [0 to 0]
  Serogroup A/H3N2 Post-vaccination 2 | 100 | 100 [0 to 0] | 99 [0 to 0] | 100 [0 to 0]
  Serogroup B Pre-vaccination | 2 | 2 [0 to 0] | 9 [0 to 0] | 3 [0 to 0]
  Serogroup B Post-vaccination 1 | 5 | 10 [0 to 0] | 47 [0 to 0] | 42 [0 to 0]
  Serogroup B Post-vaccination 2 | 44 | 21 [0 to 0] | 63 [0 to 0] | 58 [0 to 0]

4. Secondary Outcome: Percentage of Participants That Achieved Seroconversion Post-vaccination With Either a Fluzone Intradermal or a Fluzone Intramuscular Vaccine
Description: Seroconversion was defined as the conversion to a post-vaccination titer of ≥ 40 for subjects with pre-vaccination titer < 10, or at least a 4-fold increase in post vaccination titer for subjects with pre vaccination titer ≥ 10.
Time Frame: Day 28 post-vaccination
Population: Seroconversion to vaccine antigens were determined in the per-protocol population
Measure: Number; unit: Percentage of Participants
Arm/Group | Group 1: Fluzone ID at Age 6 to 35 Months | Group 2: Fluzone IM 6 to 35 Months Age Group | Group 3: Fluzone ID at 3 to 8 Years Age | Group 4: Fluzone IM 3 to 8 Years Age
Number analyzed (Participants) | 69 | 97 | 160 | 120
Percentage of Participants
  Serogroup A/H1N1 Post-vaccination 1 | 52 | 75 [0 to 0] | 65 [0 to 0] | 74 [0 to 0]
  Serogroup A/H1N1 Post-vaccination 2 | 91 | 88 [0 to 0] | 70 [0 to 0] | 78 [0 to 0]
  Serogroup A/H3N2 Post-vaccination 1 | 81 | 80 [0 to 0] | 44 [0 to 0] | 63 [0 to 0]
  Serogroup A/H3N2 Post-vaccination 2 | 88 | 91 [0 to 0] | 50 [0 to 0] | 62 [0 to 0]
  Serogroup B Post-vaccination 1 | 5 | 10 [0 to 0] | 44 [0 to 0] | 40 [0 to 0]
  Serogroup B Post-vaccination 2 | 44 | 21 [0 to 0] | 55 [0 to 0] | 53 [0 to 0]

5. Secondary Outcome: Number of Participants Reporting a Solicited Injection Site or Systemic Reactions After Each Vaccination With Either a Fluzone Intradermal or a Fluzone Intramuscular Vaccine - Age 6 to 35 Months.
Description: Solicited injection site reactions: Tenderness, Redness, Swelling, Induration and Ecchymosis. Solicited Systemic reaction: Fever (Temperature), Vomiting, Abnormal crying, Drowsiness, Loss of Appetite, and Irritability.
Time Frame: Day 0 to Day 7 post-vaccination
Population: Safety parameters were determined post-vaccination in the safety, intend-to-treat population.
Measure: Number; unit: Participants
Arm/Group | Group 1: Fluzone ID at Age 6 to 35 Months | Group 2: Fluzone IM 6 to 35 Months Age Group | Group 3: Fluzone ID at 3 to 8 Years Age | Group 4: Fluzone IM 3 to 8 Years Age
Number analyzed (Participants) | 97 | 97 | 0 | 0
Participants
  Any injection site tenderness Injection 1 | 51 | 43 |  |
  Grade 3 Tenderness (Reduced movement) | 0 | 0 |  |
  Any Injection site redness Injection 1 | 48 | 27 |  |
  Grade 3 redness ( ≥ 5 cm) | 0 | 0 |  |
  Any Injection site swelling Injection 1 | 23 | 15 |  |
  Grade 3 swelling ( ≥ 5 cm) | 0 | 0 |  |
  Any Injection site induration Injection 1 | 24 | 13 |  |
  Grade 3 induration ( ≥ 5 cm) | 0 | 0 |  |
  Any Injection site ecchymosis Injection 1 | 12 | 13 |  |
  Grade 3 ecchymosis ( ≥ 5 cm) | 1 | 0 |  |
  Any injection site tenderness Injection 2 | 48 | 49 |  |
  Grade 3 Tenderness (Reduced movement) | 1 | 1 |  |
  Any Injection site redness Injection 2 | 48 | 28 |  |
  Grade 3 redness ( ≥ 5 cm) | 1 | 0 |  |
  Any Injection site swelling Injection 2 | 18 | 13 |  |
  Grade 3 swelling ( ≥ 5 cm) | 1 | 0 |  |
  Any Injection site induration Injection 2 | 18 | 14 |  |
  Grade 3 induration ( ≥ 5 cm) | 0 | 0 |  |
  Any Injection site ecchymosis Injection 2 | 23 | 13 |  |
  Grade 3 ecchymosis ( ≥ 5 cm) | 1 | 0 |  |
  Any Solicited Fever Injection 1 | 10 | 10 |  |
  Grade 3 Fever > 103.1°F | 1 | 0 |  |
  Any Solicited Vomiting Injection 1 | 5 | 6 |  |
  Grade 3 Vomiting ≥ 6 episodes per 24 hours | 0 | 0 |  |
  Any Solicited Crying Abnormal Injection 1 | 17 | 29 |  |
  Grade 3 Crying Abnormal >3 hours | 3 | 0 |  |
  Any Solicited Drowsiness Injection 1 | 21 | 24 |  |
  Grade 3 Drowsiness Sleeping most of the time | 3 | 0 |  |
  Any Solicited Appetite Lost Injection 1 | 20 | 21 |  |
  Grade 3 Appetite Lost refuses most feeds | 3 | 0 |  |
  Any Solicited Irritability Injection 1 | 37 | 39 |  |
  Grade 3 Irritability inconsolable | 2 | 1 |  |
  Any Solicited Fever Injection 2 | 6 | 9 |  |
  Grade 3 Fever > 103.1°F | 0 | 1 |  |
  Any Solicited Vomiting Injection 2 | 4 | 7 |  |
  Grade 3 Vomiting ≥ 6 episodes per 24 hours | 0 | 0 |  |
  Any Solicited Crying Abnormal Injection 2 | 19 | 16 |  |
  Grade 3 Crying Abnormal >3 hours | 1 | 2 |  |
  Any Solicited Drowsiness Injection 2 | 13 | 23 |  |
  Grade 3 Drowsiness Sleeping most of the time | 0 | 0 |  |
  Any Solicited Appetite Lost Injection 2 | 18 | 17 |  |
  Grade 3 Appetite Lost refuses most feeds | 1 | 1 |  |
  Any Solicited Irritability Injection 2 | 30 | 30 |  |
  Grade 3 Irritability inconsolable | 3 | 4 |  |

6. Secondary Outcome: Number of Participants Reporting a Solicited Injection Site or Systemic Reactions After Each Vaccination With Either a Fluzone Intradermal or a Fluzone Intramuscular Vaccine - Age 3 to 8 Year Olds
Description: Solicited injection site reactions: Pain, Redness, Swelling, Induration and Ecchymosis. Solicited Systemic reaction: Fever (Temperature), Headache, Malaise, and Myalgia.
Time Frame: Day 0 to Day 7 post-vaccination
Population: Safety parameters were determined post-vaccination in the safety, intend-to-treat population.
Measure: Number; unit: Participants
Arm/Group | Group 1: Fluzone ID at Age 6 to 35 Months | Group 2: Fluzone IM 6 to 35 Months Age Group | Group 3: Fluzone ID at 3 to 8 Years Age | Group 4: Fluzone IM 3 to 8 Years Age
Number analyzed (Participants) | 0 | 0 | 160 | 163
Participants
  Any injection site Pain Injection 1 |  |  | 93 | 89
  Grade 3 Pain (Reduced movement) |  |  | 0 | 0
  Any Injection site Redness Injection 1 |  |  | 98 | 42
  Grade 3 Redness ( ≥ 5 cm) |  |  | 2 | 1
  Any Injection site Swelling Injection 1 |  |  | 59 | 30
  Grade 3 Swelling ( ≥ 5 cm) |  |  | 1 | 0
  Any Injection site Induration Injection 1 |  |  | 56 | 25
  Grade 3 Induration ( ≥ 5 cm) |  |  | 1 | 0
  Any Injection site Ecchymosis Injection 1 |  |  | 18 | 19
  Grade 3 Ecchymosis ( ≥ 5 cm) |  |  | 0 | 1
  Any Solicited Pruritus Injection 1 |  |  | 23 | 11
  Any injection site pain Injection 2 |  |  | 98 | 90
  Grade 3 Pain (Reduced movement) |  |  | 0 | 1
  Any Injection site Redness Injection 2 |  |  | 94 | 40
  Grade 3 Redness (≥ 5 cm) |  |  | 1 | 1
  Any Injection site Swelling Injection 2 |  |  | 61 | 21
  Grade 3 swelling ( ≥ 5 cm) |  |  | 1 | 0
  Any Injection site Induration Injection 2 |  |  | 50 | 17
  Grade 3 Induration (≥ 5 cm) |  |  | 1 | 0
  Any Injection site Ecchymosis Injection 2 |  |  | 18 | 22
  Grade 3 Ecchymosis (≥ 5 cm) |  |  | 0 | 0
  Any Solicited Pruritus Injection 2 |  |  | 15 | 19
  Any Solicited Fever Injection 1 |  |  | 10 | 18
  Grade 3 Fever > 102.2°F |  |  | 2 | 3
  Any Solicited Headache Injection 1 |  |  | 22 | 25
  Grade 3 Headache Prevents daily activities |  |  | 1 | 1
  Any Solicited Malaise Injection 1 |  |  | 21 | 30
  Grade 3 Malaise Prevents daily activities |  |  | 1 | 2
  Any Solicited Myalgia Injection 1 |  |  | 24 | 42
  Grade 3 Myalgia Prevents daily activities |  |  | 0 | 0
  Any Solicited Fever Injection 2 |  |  | 16 | 14
  Grade 3 Fever > 102.2°F |  |  | 0 | 2
  Any Solicited Headache Injection 2 |  |  | 15 | 17
  Grade 3 Headache Prevents daily activities |  |  | 2 | 2
  Any Solicited Malaise Injection 2 |  |  | 24 | 21
  Grade 3 Malaise Prevents daily activities |  |  | 1 | 1
  Any Solicited Myalgia Injection 2 |  |  | 24 | 25
  Grade 3 Myalgia Prevents daily activities |  |  | 2 | 0

ADVERSE EVENTS:
Time Frame: Adverse events data were collected from the day of vaccination to up to 6 months post-vaccination 2
Arm/Group | Group 1: Fluzone ID at Age 6 to 35 Months | Group 2: Fluzone IM 6 to 35 Months Age Group | Group 3: Fluzone ID at 3 to 8 Years Age | Group 4: Fluzone IM 3 to 8 Years Age
Serious Adverse Events (participants affected / at risk) | 1/97 | 1/97 | 1/160 | 1/163
Other Adverse Events (participants affected / at risk) | 51/97 | 49/97 | 98/160 | 90/163
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group 1: Fluzone ID at Age 6 to 35 Months (N=97) | Group 2: Fluzone IM 6 to 35 Months Age Group (N=97) | Group 3: Fluzone ID at 3 to 8 Years Age (N=160) | Group 4: Fluzone IM 3 to 8 Years Age (N=163)
Gastroenteritis viral (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Viral infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Autism (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5.00% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Group 1: Fluzone ID at Age 6 to 35 Months (N=97) | Group 2: Fluzone IM 6 to 35 Months Age Group (N=97) | Group 3: Fluzone ID at 3 to 8 Years Age (N=160) | Group 4: Fluzone IM 3 to 8 Years Age (N=163)
Conjunctivitis (Eye disorders) | 5 (5) | 6 (6) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 7 (8) | 9 (9) | 15 (15) | 3 (3)
Teething (Gastrointestinal disorders) | 7 (8) | 6 (11) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 3 (3) | 6 (6) | 14 (14) | 12 (13)
Pyrexia (General disorders) | 8 (9) | 22 (27) | 13 (13) | 14 (14)
Vessel puncture site bruise (General disorders) | 11 (12) | 15 (17) | 11 (11) | 16 (19)
Bronchitis (Infections and infestations) | 0 (0) | 5 (5) | 0 (0) | 0 (0)
Croup infections (Infections and infestations) | 4 (4) | 5 (5) | 4 (4) | 3 (4)
Gastroenteritis (Infections and infestations) | 5 (5) | 0 (0) | 4 (4) | 2 (2)
Nasopharyngitis (Infections and infestations) | 14 (16) | 9 (11) | 4 (5) | 18 (20)
Otitis media (Infections and infestations) | 17 (19) | 23 (27) | 8 (9) | 8 (8)
Sinusitis (Infections and infestations) | 4 (4) | 7 (7) | 5 (5) | 4 (4)
Upper respiratory tract infection (Infections and infestations) | 15 (17) | 18 (23) | 9 (10) | 7 (10)
Viral infection (Infections and infestations) | 2 (2) | 5 (5) | 5 (5) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 33 (44) | 32 (39) | 46 (60) | 42 (55)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 7 (11) | 4 (6) | 4 (5) | 9 (11)
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 7 (8) | 12 (15)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 18 (24) | 19 (26) | 19 (30) | 20 (26)
Injection site Tenderness (General disorders) | 51/93 (51) | 49/87 (49) | 98/137 (98) | 90/145 (90)
Injection site Redness (General disorders) | 48/93 (48) | 28/87 (28) | 98/143 (98) | 42/151 (42)
Injection site Swelling (General disorders) | 23/88 (23) | 15/90 (15) | 61/137 (61) | 30/151 (30)
Injection site Induration (General disorders) | 24/93 (24) | 14/87 (14) | 56/143 (56) | 25/151 (25)
Injection site Ecchymosis (General disorders) | 23/88 (23) | 13/87 (13) | 18/143 (18) | 22/145 (22)
Vomiting (Gastrointestinal disorders) | 5/93 (5) | 7/86 (7) | 0 | 0
Crying abnormal (Psychiatric disorders) | 17/93 (17) | 29/91 (29) | 0 | 0
Drowsiness (Nervous system disorders) | 21/93 (21) | 24/91 (24) | 0 | 0
Appetite lost (Gastrointestinal disorders) | 20/93 (20) | 21/91 (21) | 0 | 0
Irritability (Nervous system disorders) | 37/93 (37) | 39/91 (39) | 0 | 0
Malaise (General disorders) | 0 | 0 | 24/136 (24) | 30/150 (30)
Myalgia (General disorders) | 0 | 0 | 24/141 (24) | 42/150 (42)
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 23/139 (23) | 19/144 (19)
Headache (Nervous system disorders) | 0 | 0 | 22/141 (22) | 25/150 (25)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor must have the opportunity to review at least 60 days prior to submission for publication or presentation. If review indicates that potentially patentable subject matter would be disclosed, publication or public disclosure may be delayed for a maximum of an additional 60 days to allow for filing the necessary patent applications.